CLINICAL TRIAL: NCT00787085
Title: The Significance of Funguria in Hospitalized Patients (FACES)
Brief Title: The Significance of Funguria in Hospitalized Patients
Acronym: FACES
Status: Completed | Type: Observational
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Cedars-Sinai Medical Center (Other)
Responsible Party: Loren Gregory Miller, M.D., M.P.H., Principal Investigator, Los Angeles Biomedical Research Institute
Other Study IDs: 10024-05; NIH-AI01831
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Urinary Tract Infections
Keywords: Funguria; Epidemiology; Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood cultures
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case: Patients hospitalized with a urine or blood culture positive for fungi
- Control: Patients hospitalized with a urine culture negative for fungi

SUMMARY:
This investigation is a epidemiologic case-control study of the risk factors associated with nosocomial funguria (fungi in the urine).

DETAILED DESCRIPTION:
A recent large multi-center national surveillance survey of almost 5000 nosocomial (hospital based) urine isolates from medical intensive care units demonstrated that fungi comprised nearly 40% of urine isolates. Little is known about distinguishing fungi that cause colonization from those causing infection.

The objective of this study is to define the epidemiology of nosocomial funguria and natural history of patients that develop funguria while hospitalized.

Patients who may have eligible for this study will be identified from microbiology laboratory specimens at the Harbor-UCLA Medical Center and Cedars-Sinai Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at least 12 hours of any age (< 1 day to > 100 years of age) AND a urine or blood culture positive for fungi, OR urine culture negative for fungi (control group)

Exclusion Criteria:

* Patients already surveyed for funguria during current hospitalization and patients already being followed for recognized funguria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized at the Harbor-UCLA Medical Center and Cedars-Sinai Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 919 (Actual)
Dates: Start 2001-09; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Funguria | Hospitalization day 0, 3, 7, 14, and every 7 days thereafter until hospital discharge or death

CONTACTS AND LOCATIONS:
Overall Officials: Loren G Miller, M.D., M.P.H., Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (2):
- United States (2):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California